CLINICAL TRIAL: NCT01315041
Title: Effects of Homeopathic Medicine "Pi" on Hot Flushes of Women With Menopausal Symptoms
Brief Title: "Pi" and Hot Flushes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Casa Espirita Terra de Ismael (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fabio Carmona, Assistant Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pi2011
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Menopausal Symptom Relief
MeSH Terms: interventions — Homeopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Pi" medicine (Active Comparator)
  Interventions: Drug: Capsicum frutescens fruits, homeopathic medicine
- Placebo (Placebo Comparator)
  Interventions: Drug: Inert alcoholic solution

INTERVENTIONS:
Drug: Capsicum frutescens fruits, homeopathic medicine — 5 drops, PO, 3 times a day, during 16 weeks
  Arms: "Pi" medicine
Drug: Inert alcoholic solution — 5 drops, PO, 3 times a day, during 16 weeks
  Arms: Placebo

SUMMARY:
Hot flushes are common symptoms in women after menopause, and are important causes of discomfort and lead to high number of medical consultations. Hormone replacement therapy is an effective treatment, however it can bring undesirable consequences and may be contraindicated for some women. Options are inhibitors of serotonin or serotonin-norepinephrine reuptake, gabapentin, herbal medicines and homeopathy. None of these therapies is widely accepted of effective. Therefore, the search for new therapeutic options is highly desirable. Ingestion of malagueta pepper fruits (Capsicum frutescens L. var. malagueta) causes sensations similar to those experienced by menopausal women during hot flushes. By the principle of homeopathy, "the like cures the like", the objectives of this study are: (a) to determinate whether pathogenesis of a homeopathic medicine made from C. frutescens fruits include symptoms like hot flushes, and (b) whether this medicine is effective on hot flushes relief in women after menopause. There will be 2 distinct phases. Phase 1 is the determination of the medicine's pathogenesis in healthy volunteers, in a randomized placebo-controlled, double-blind design. Phase 2 is the investigation of the medicine's effects on hot flushes of women after menopause, in a randomized placebo-controlled, double-blind design. The investigators expect a significant reduction on symptoms perception, assessed by internationally validated tools. The study is expected to last for 18 months, with 36 patients included in each phase.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1: healthy volunteers
* Phase 2: menopaused women with hot flushes

Exclusion Criteria:

* Illiteracy;
* Have been enrolled in another clinical trial within the last 6 months;
* Use of pharmacological therapies for hot flushes;
* Have any degree of vulnerability;
* Allergy or hypersensitivity to Capsicum species;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
MYMOP (Measure Yourself Medical Outcome Profile) | 4 and 16 weeks
ORIDL (Outcome Related to Impact on Daily Living) | 4 and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Carmona, MD, PhD, Study Director — University of Sao Paulo; Mateus A Angelucci, MD, MSc, Principal Investigator — University of Sao Paulo; Ana MS Pereira, PhD, Study Chair — University of Ribeirao Preto; Edson Z Martinez, PhD, Study Director — University of Sao Paulo
Locations (1):
- Casa Espirita Terra de Ismael, Jardinópolis, São Paulo, Brazil